CLINICAL TRIAL: NCT05321511
Title: Double Ovarian Stimulation (DuoStim) Comparison of Triggers: Is There Any Advantage Using 3 Different Methods of Trigger for the Second Egg Collection in Predicted Low Responders?
Brief Title: Comparison of Triggers in Double Ovarian Stimulation (DuoStim).
Acronym: COTRID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Andrea Bernabeu García, Co-Director, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB-0121
Record Dates: First submitted 2022-03-24; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: IVF; LOW OVARIAN RESPONSE
MeSH Terms: interventions — Triptorelin Pamoate; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- a-GnRH (Active Comparator): Administration of triptorelin acetate 0.2 mg for final oocyte maturation.
  Interventions: Drug: Triptorelin acetate (a-GnRH)
- hCG (Active Comparator): Administration of coriogonadotropine alfa 250 mcg for final oocyte maturation.
  Interventions: Drug: Ovitrelle® (hCG)
- a-GnRH + hCG (Experimental): Administration of triptorelin acetate 0.2 mg and coriogonadotropine alfa 250 mcg for final oocyte maturation.
  Interventions: Drug: Decapeptyl 0.1 mg® (a-GnRH) and Ovitrelle® (hCG) used together

INTERVENTIONS:
Drug: Triptorelin acetate (a-GnRH) — Adminsitration of triptoreline acetate 0.2 mg for final oocyte maturation in the second ovarian stimuation inthe Double stimulation protocol.
  Other Names: Decapeptyl 0.1 mg®
  Arms: a-GnRH
Drug: Ovitrelle® (hCG) — Adminsitration of coriogonadotropine alfa 250 mcg for final oocyte maturation in the second ovarian stimuation inthe Double stimulation protocol.
  Arms: hCG
Drug: Decapeptyl 0.1 mg® (a-GnRH) and Ovitrelle® (hCG) used together — Adminsitration of triptoreline acetate 0.2 mg and coriogonadotropine alfa 250 mcg for final oocyte maturation in the second ovarian stimuation inthe Double stimulation protocol.
  Arms: a-GnRH + hCG

SUMMARY:
This study aims to investigate the efficacy of 3 different trigggers used for final maturation in the second ovarian stimulation in double stimulation protocol (aGnRH and hCG-rec vs. aGnRH only vs. hCG-rec only). The main objective is to compare the number of all retrieved oocytes and mature oocytes in patients predicted to be low ovarian responders.

This is a controlled randomized clinical study where 165 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* BMI below 32
* Presence of both ovaries
* Indication for ovarian stimulation under Double Stimulation protocol (Duo Stim)
* Meeting the criteria for Duo Stim
* Medical history, history and physical examination without alterations
* AMH and AFV results in accordnace to Poseidon classification group 3 or 4 no more than 6 months prior to signing the consent form
* Ability to participate and comply with the study protocol.
* To have given written consent
* Normal karyotype and fragile X.

Exclusion Criteria:

* Non-compliance with instructions and/or non-formalization of consents or legal requirements for IVF.
* Concurrent participation in another study

Ages: 28 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
number of retrieved oocytes | through study completion, usually will be evaluated on the last day of the treatment
  number of oocytes retrieved in the second ovarian stimulation in the double stimulation protocol.
number of mature (MII) oocytes | through study completion, usually will be evaluated on the last day of the treatment
  number of mature (MII) oocytes retrieved in the second ovarian stimulation in the double stimulation protocol.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Instituto Bernabeu, Palma de Mallorca, Mallorca
  - Instituto Bernabeu, Albacete
  - Instituto Bernabeu, Alicante
  - Instituto Bernabeu, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castillo JC, Haahr T, Martinez-Moya M, Humaidan P. Gonadotropin-releasing hormone agonist ovulation trigger-beyond OHSS prevention. Ups J Med Sci. 2020 May;125(2):138-143. doi: 10.1080/03009734.2020.1737599. Epub 2020 Mar 25. PMID 32208810
- [Result] Pereira N, Elias RT, Neri QV, Gerber RS, Lekovich JP, Palermo GD, Rosenwaks Z. Adjuvant gonadotrophin-releasing hormone agonist trigger with human chorionic gonadotrophin to enhance ooplasmic maturity. Reprod Biomed Online. 2016 Nov;33(5):568-574. doi: 10.1016/j.rbmo.2016.08.009. Epub 2016 Aug 20. PMID 27567429
- [Result] Moffat R, Pirtea P, Gayet V, Wolf JP, Chapron C, de Ziegler D. Dual ovarian stimulation is a new viable option for enhancing the oocyte yield when the time for assisted reproductive technnology is limited. Reprod Biomed Online. 2014 Dec;29(6):659-61. doi: 10.1016/j.rbmo.2014.08.010. Epub 2014 Sep 4. PMID 25311972
- [Result] Lin MH, Wu FS, Hwu YM, Lee RK, Li RS, Li SH. Dual trigger with gonadotropin releasing hormone agonist and human chorionic gonadotropin significantly improves live birth rate for women with diminished ovarian reserve. Reprod Biol Endocrinol. 2019 Jan 4;17(1):7. doi: 10.1186/s12958-018-0451-x. PMID 30609935
- [Result] Haas J, Zilberberg E, Dar S, Kedem A, Machtinger R, Orvieto R. Co-administration of GnRH-agonist and hCG for final oocyte maturation (double trigger) in patients with low number of oocytes retrieved per number of preovulatory follicles--a preliminary report. J Ovarian Res. 2014 Aug 2;7:77. doi: 10.1186/1757-2215-7-77. PMID 25296696
- [Result] Zhang J, Wang Y, Mao X, Chen Q, Hong Q, Cai R, Zhang S, Kuang Y. Dual trigger of final oocyte maturation in poor ovarian responders undergoing IVF/ICSI cycles. Reprod Biomed Online. 2017 Dec;35(6):701-707. doi: 10.1016/j.rbmo.2017.09.002. Epub 2017 Sep 21. PMID 28993105